CLINICAL TRIAL: NCT02130466
Title: A Phase I/II Study to Assess the Safety and Efficacy of MK-3475 in Combination With Trametinib and Dabrafenib in Subjects With Advanced Melanoma
Brief Title: A Study of the Safety and Efficacy of Pembrolizumab (MK-3475) in Combination With Trametinib and Dabrafenib in Participants With Advanced Melanoma (MK-3475-022/KEYNOTE-022)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-022; MK-3475-022 (Other: Merck); KEYNOTE-022 (Other: Merck); 2015-000681-55 (EudraCT Number)
Expanded Access: NCT02083484 (No longer available)
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-06

CONDITIONS: Melanoma; Solid Tumors
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; dabrafenib; trametinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part 1:pembrolizumab 2 mg/kg+dabrafenib150 mg+trametinib 2 mg (Experimental): Participants with BRAF mutant melanoma received 2 mg/kg pembrolizumab administered by intravenous (IV) infusion on Days 1 and 22 of each 6-week cycle (Q6W); 150 mg/day total dabrafenib orally, in a divided dose, twice a day (BID) starting on Day 1 and continuing up until study treatment discontinuation; and 2 mg trametinib orally once a day (QD) starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Dabrafenib; Drug: Trametinib
- Part 1:pembrolizumab 2 mg/kg+trametinib 2 mg (Experimental): Participants with BRAF wild-type melanoma received 2 mg/kg pembrolizumab administered by IV infusion on Days 1 and 22 Q6W and 2 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 1:pembrolizumab 2 mg/kg+trametinib 1.5 mg (Experimental): Participants with BRAF wild-type melanoma received 2 mg/kg pembrolizumab administered by IV infusion on Days 1 and 22 Q6W and 1.5 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 2:pembrolizumab 2 mg/kg+dabrafenib 150 mg+trametinib 2 mg (Experimental): Participants with BRAF mutant melanoma received 2 mg/kg pembrolizumab administered by IV infusion on Days 1 and 22 Q6W; 150 mg/day total dabrafenib orally, in a divided dose, BID starting on Day 1 and continuing up until study treatment discontinuation; and 2 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Dabrafenib; Drug: Trametinib
- Part 2:pembrolizumab 2 mg/kg+trametinib 1.5 mg (Experimental): Participants with BRAF wild-type melanoma received 2 mg/kg pembrolizumab administered by IV infusion on Days 1 and 22 Q6W and 1.5 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 3:pembrolizumab 2 mg/kg+dabrafenib 150 mg+trametinib 2 mg (Experimental): Participants with BRAF mutant melanoma received 2 mg/kg pembrolizumab administered by IV infusion on Days 1 and 22 Q6W; 150 mg/day total dabrafenib orally, in a divided dose, BID starting on Day 1 and continuing up until study treatment discontinuation; and 2 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Dabrafenib; Drug: Trametinib
- Part 3:placebo+dabrafenib 150 mg+trametinib 2 mg (Placebo Comparator): Participants with BRAF mutant melanoma received saline placebo administered by IV infusion on Days 1 and 22 Q6W; 150 mg/day total dabrafenib orally, in a divided dose, BID starting on Day 1 and continuing up until study treatment discontinuation; and 2 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Placebo
- Part 4:trametinib 2 mg for 4 weeks+pembrolizumab 200 mg+trametinib 2 mg concurrent dosing (Experimental): Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 2 mg trametinib orally QD for 4 weeks. Starting with Week 5, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 of each 3-week cycle (Q3W) and a concurrent dosing schedule of 2 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 4:trametinib 1.5 mg for 2 weeks+pembrolizumab 200 mg+trametinib 1.5 mg concurrent dosing (Experimental): Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 1.5 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and a concurrent dosing schedule of 1.5 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 4:trametinib 1.5 mg for 4 weeks+pembrolizumab 200 mg+trametinib 1.5 mg concurrent dosing (Experimental): Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 1.5 mg trametinib orally QD for 4 weeks. Starting with Week 5, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and a concurrent dosing schedule of 1.5 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 4:trametinib 2 mg for 2 weeks+pembrolizumab 200 mg+trametinib 2 mg intermittent dosing (Experimental): Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 2 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent dose schedule of 2 mg trametinib orally QD with 1 week OFF trametinib and 2 weeks ON trametinib continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 4:trametinib 1.5 mg for 2 weeks+pembrolizumab 200 mg+trametinib 1.5 mg intermittent dosing (Experimental): Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 1.5 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent dose schedule of 1.5 mg trametinib orally QD with 1 week OFF trametinib and 2 weeks ON trametinib continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 5:trametinib 1.5 mg for 2 weeks+pembrolizumab 200 mg+trametinib 1.5 mg concurrent dosing (Experimental): Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 1.5 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and a concurrent dosing schedule of 1.5 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Part 5:trametinib 2 mg for 2 weeks+pembrolizumab 200 mg+trametinib 2 mg intermittent dosing (Experimental): Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 2 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent dose schedule of 2 mg trametinib orally QD with 1 week OFF trametinib and 2 weeks ON trametinib continuing up until study treatment discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Part 1:pembrolizumab 2 mg/kg+dabrafenib150 mg+trametinib 2 mg; Part 1:pembrolizumab 2 mg/kg+trametinib 1.5 mg; Part 1:pembrolizumab 2 mg/kg+trametinib 2 mg; Part 2:pembrolizumab 2 mg/kg+dabrafenib 150 mg+trametinib 2 mg; Part 2:pembrolizumab 2 mg/kg+trametinib 1.5 mg; Part 3:pembrolizumab 2 mg/kg+dabrafenib 150 mg+trametinib 2 mg; Part 4:trametinib 1.5 mg for 2 weeks+pembrolizumab 200 mg+trametinib 1.5 mg concurrent dosing; Part 4:trametinib 1.5 mg for 2 weeks+pembrolizumab 200 mg+trametinib 1.5 mg intermittent dosing; Part 4:trametinib 1.5 mg for 4 weeks+pembrolizumab 200 mg+trametinib 1.5 mg concurrent dosing; Part 4:trametinib 2 mg for 2 weeks+pembrolizumab 200 mg+trametinib 2 mg intermittent dosing; Part 4:trametinib 2 mg for 4 weeks+pembrolizumab 200 mg+trametinib 2 mg concurrent dosing; Part 5:trametinib 1.5 mg for 2 weeks+pembrolizumab 200 mg+trametinib 1.5 mg concurrent dosing; Part 5:trametinib 2 mg for 2 weeks+pembrolizumab 200 mg+trametinib 2 mg intermittent dosing
Drug: Dabrafenib — oral capsule
  Other Names: TAFINLAR®
  Arms: Part 1:pembrolizumab 2 mg/kg+dabrafenib150 mg+trametinib 2 mg; Part 2:pembrolizumab 2 mg/kg+dabrafenib 150 mg+trametinib 2 mg; Part 3:pembrolizumab 2 mg/kg+dabrafenib 150 mg+trametinib 2 mg; Part 3:placebo+dabrafenib 150 mg+trametinib 2 mg
Drug: Trametinib — oral tablet
  Other Names: MEKINIST®
Drug: Placebo — IV infusion
  Arms: Part 3:placebo+dabrafenib 150 mg+trametinib 2 mg

SUMMARY:
This is a 5-part dose-finding and preliminary efficacy study of pembrolizumab (Pembro) + dabrafenib (D) + trametinib (T) for participants with advanced melanoma and solid tumors.

Parts 1 and 2 are open-label to find and confirm the maximum tolerated dose (MTD)/maximum administered dose (MAD) for Pembro+D+T. The primary hypothesis (Parts 1 and 2) is that Pembro+D+T is sufficiently well-tolerated to permit clinical investigation.

Part 3 is a double-blind study of Pembro+D+T versus placebo+D+T. The primary study hypothesis (Part 3 only) is that the Pembro+D+T improves progression-free survival (PFS) compared with placebo+D+T.

Part 4 is nonrandomized and open-label and is designed to evaluate the safety and tolerability and identify the MTD or MAD of Pembro+T in participants who have v-raf murine sarcoma viral oncogene homolog B1 [BRAF] mutation-negative (without V600 E or K) melanoma or solid tumors [irrespective of BRAF status]. The primary hypothesis (Part 4) is that Pembro+T is sufficiently well-tolerated to permit clinical investigation.

Part 5 will confirm the dose(s) identified in Part 4 in participants BRAF wild type [without V600E or K] melanoma or solid tumors [irrespective of BRAF status] and will further evaluate the safety and preliminary efficacy (Objective Response Rate [ORR]) of Pembro+T in participants who have BRAF wild type [without V600E or K] melanoma or solid tumors [irrespective of BRAF status]. The primary hypotheses (Part 5) are that Pembro+T is sufficiently well-tolerated at the MTD/MAD to permit further clinical investigation and is effective in attaining objective responses based upon Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator review in participants who have melanoma without BRAF V600 E or K mutations. With Amendment 5 (21-Mar-2019), the Part 5 expansion cohort will not be pursued following the completion of Part 5 dose confirmation.

Parts 1 and 2 of the study may also explore, if needed based on tolerability, the backup combinations of open-label Pembro+T (for BRAF mutation-negative participants) or Pembro+D (for BRAF mutation-positive participants). These will run concurrently with the Pembro+D+T arm.

ELIGIBILITY:
Inclusion criteria:

* Histologically-confirmed diagnosis of advanced (unresectable Stage III) or metastatic (Stage IV) melanoma excluding mucosal, or ocular melanoma (or a histologically or cytologically-documented locally-advanced or metastatic solid malignancy in Parts 4 and 5)
* At least 1 measurable lesion as defined by RECIST 1.1 on imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI])
* For solid tumors other than melanoma, (in Part 4 or 5 [dose confirmation only]), participants must have a malignancy that is incurable and has either: (a) failed prior standard therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate by the participants and treating physician. There is no limit to the number of prior treatment regimens, but prior treatment(s) should not include compounds targeting programmed cell death 1 (PD-1), programmed cell death ligand 1 (PD-L1), BRAF, or mitogen-activated protein kinase (MEK). Treatment must end at least 4 weeks prior to randomization
* BRAF mutation-positive (V600 E or K) melanoma for Parts 1, 2 and 3, or for Parts 1, 2, 4 and 5 only BRAF mutation-negative (wild type) melanoma with documented progression of ≥1 measurable lesion after prior therapy (if prior therapy was received). The inclusion criterion does not apply to participants with solid tumors in Parts 4 and 5 (dose confirmation only)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Anticipated life expectancy of at least 3 months
* Able to swallow and retain oral medication and no clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Adequate organ function
* Provide tissue for biomarker analysis from a newly or recently-obtained biopsy (within 90 days of Study Day 1) of a tumor lesion not previously irradiated
* Female participants of non-childbearing potential must be willing to use highly effective contraceptive measures from the Screening Visit (Visit 1) through 120 days after the last dose of study drug; male participants must agree to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug
* Female participants of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study drug

Exclusion criteria:

* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study drug
* Prior systemic therapy (for participants who are BRAF mutation-positive), or BRAF mutation-negative and has received >1 prior systemic therapy for metastatic melanoma
* Prior therapy with compounds targeting PD-1, PD-L1, BRAF, MEK or other molecules in the mitogen-activated protein kinase (MAPK) pathway
* BRAF mutation-positive and has received prior systemic therapy with ipilimumab or other anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) blocking antibodies. The BRAF exclusion criterion does not apply to participants with solid tumor in Parts 4 and 5 (dose confirmation only)
* Chemotherapy, radioactive, or biological cancer therapy within 4 weeks prior to the first dose of study drug, or not recovered from clinically significant adverse events due to cancer therapeutics administered more than 4 weeks prior to the first dose of study drug
* Expected to require any other form of systemic or localized antineoplastic therapy while in this study
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include early stage cancers (carcinoma in situ or stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active infection requiring systemic therapy
* Active autoimmune disease, or documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents
* Previous severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
* On chronic systemic steroid therapy (>10 mg/day prednisone or equivalent) within 2 weeks prior to first dose of study drug or on any other form of immunosuppressive medication
* History or evidence of cardiovascular risk
* Uncorrectable electrolyte abnormalities, long QT syndrome or taking medications known to prolong the QT interval
* History of prior or current retinal vein occlusion (RVO)
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs, their excipients, and/or dimethyl sulfoxide (DMSO)
* Has had an allogeneic tissue/solid organ transplant, prior stem cell or bone marrow transplant
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Human immunodeficiency virus (HIV)
* Hepatitis B or C
* Received a live vaccine within 30 days prior to first dose of study drug
* Pregnant or breastfeeding or expecting to conceive or father children from the Screening Visit (Visit 1) through 120 days after last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ribas A, Lawrence D, Atkinson V, Agarwal S, Miller WH Jr, Carlino MS, Fisher R, Long GV, Hodi FS, Tsoi J, Grasso CS, Mookerjee B, Zhao Q, Ghori R, Moreno BH, Ibrahim N, Hamid O. Combined BRAF and MEK inhibition with PD-1 blockade immunotherapy in BRAF-mutant melanoma. Nat Med. 2019 Jun;25(6):936-940. doi: 10.1038/s41591-019-0476-5. Epub 2019 Jun 6. PMID 31171879
- [Result] Ascierto PA, Ferrucci PF, Fisher R, Del Vecchio M, Atkinson V, Schmidt H, Schachter J, Queirolo P, Long GV, Di Giacomo AM, Svane IM, Lotem M, Bar-Sela G, Couture F, Mookerjee B, Ghori R, Ibrahim N, Moreno BH, Ribas A. Dabrafenib, trametinib and pembrolizumab or placebo in BRAF-mutant melanoma. Nat Med. 2019 Jun;25(6):941-946. doi: 10.1038/s41591-019-0448-9. Epub 2019 Jun 6. PMID 31171878
- [Derived] Maio M, Carlino MS, Joshua AM, McWhirter E, Ribas A, Ascierto PA, Miller WH Jr, Butler MO, Ferrucci PF, Zielinski RR, Del Vecchio M, Gasal E, Ghori R, Diede SJ, Croydon E, Hamid O. KEYNOTE-022: Pembrolizumab with trametinib in patients with BRAF wild-type melanoma or advanced solid tumours irrespective of BRAF mutation. Eur J Cancer. 2022 Jan;160:1-11. doi: 10.1016/j.ejca.2021.09.024. Epub 2021 Nov 17. PMID 34801354
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For Parts 1 and 2 of the study the optional pembrolizumab+trametinib arm was added to the study but the optional pembrolizumab+dabrafenib arm was not implemented.
Groups:
- Part 1:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg: Participants with BRAF mutant melanoma received 2 mg/kg pembrolizumab administered by intravenous (IV) infusion on Days 1 and 22 of each 6-week cycle (Q6W); 150 mg/day total dabrafenib orally, in a divided dose, twice a day (BID) starting on Day 1 and continuing up until study treatment discontinuation; and 2 mg trametinib orally once a day (QD) starting on Day 1 and continuing up until study treatment discontinuation.
- Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg: Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 2 mg trametinib orally QD for 4 weeks. Starting with Week 5, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 of each 3-week cycle (Q3W) and a concurrent dosing schedule of 2 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
- Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg; Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg: Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 1.5 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and a concurrent dosing schedule of 1.5 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
- Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg: Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 1.5 mg trametinib orally QD for 4 weeks. Starting with Week 5, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and a concurrent dosing schedule of 1.5 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
- Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent; Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent: Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 2 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent dose schedule of 2 mg trametinib orally QD with 1 week OFF trametinib and 2 weeks ON trametinib continuing up until study treatment discontinuation.
- Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent: Participants with BRAF wild-type melanoma or solid tumors (irrespective of BRAF status) received 1.5 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent dose schedule of 1.5 mg trametinib orally QD with 1 week OFF trametinib and 2 weeks ON trametinib continuing up until study treatment discontinuation.
Period: Overall Study
Arm/Group | Part 1:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg | Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent
Started | 7 | 3 | 2 | 8 | 2 | 60 | 60 | 3 | 4 | 5 | 6 | 3 | 12 | 9
Treated | 7 | 3 | 2 | 8 | 2 | 60 | 60 | 3 | 4 | 5 | 6 | 3 | 12 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 3 | 2 | 8 | 2 | 60 | 60 | 3 | 4 | 5 | 6 | 3 | 12 | 9
Not completed — Death | 4 | 1 | 1 | 3 | 2 | 30 | 45 | 2 | 3 | 4 | 5 | 3 | 11 | 7
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participation in Study Discontinued by Sponsor | 1 | 2 | 1 | 5 | 0 | 27 | 14 | 1 | 0 | 1 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received ≥1 dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg | Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent | Total
Number analyzed (Participants) | 7 | 3 | 2 | 8 | 2 | 60 | 60 | 3 | 4 | 5 | 6 | 3 | 12 | 9 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (14.0) | 54.0 (15.7) | 68.0 (2.8) | 42.0 (14.2) | 83.0 (5.7) | 55.3 (12.0) | 57.2 (14.6) | 47.3 (19.9) | 50.0 (18.0) | 57.0 (18.0) | 55.5 (17.9) | 58.0 (12.2) | 55.7 (14.1) | 55.9 (13.3) | 55.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 5 | 0 | 27 | 24 | 0 | 2 | 3 | 5 | 2 | 8 | 6 | 86
  Male | 4 | 3 | 1 | 3 | 2 | 33 | 36 | 3 | 2 | 2 | 1 | 1 | 4 | 3 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 7 | 3 | 2 | 7 | 2 | 57 | 57 | 3 | 2 | 2 | 4 | 2 | 12 | 9 | 169
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 3 | 2 | 8 | 2 | 60 | 59 | 2 | 4 | 5 | 5 | 2 | 11 | 9 | 179
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRAF Mutation Status [Count of Participants; unit: Participants] — BRAF mutation testing was required for study inclusion and was done using methodology that detects both V600E and V600K mutations. Tumors that were BRAF mutation positive (V600 E or K) were eligible for treatment with pembrolizumab + trametinib + dabrafenib or trametinib + dabrafenib. Tumors that were BRAF mutation negative (wild type) were eligible for treatment with pembrolizumab + trametinib.
  Participants
    Mutant (BRAF Positive) | 7 | 0 | 0 | 8 | 0 | 60 | 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 135
    Wild Type (BRAF Negative) | 0 | 3 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 5 | 5 | 22
    Undetermined | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 6 | 1 | 12
    Data Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 2 | 1 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Parts 1, 2, 4, and 5: Number of Participants Who Experienced Dose-limiting Toxicities (DLTs)
Description: DLTs were graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Events were considered a DLT if occurred during the DLT evaluation period and met ≥1 of the following: significant hematologic toxicity; significant Grade ≥3 non-hematologic toxicity not previously identified or known to occur and cannot be controlled with routine supportive measures; drug-related toxicity that results in an interruption of any component of study therapy for >21 consecutive days and cannot be controlled ≤2 weeks from onset; any other Grade ≥2 non-hematological toxicity that is dose limiting with some exceptions; and liver chemistries meeting study stopping guidelines. The DLT evaluable population included all participants in Parts 1, 2, 4, and 5 who received ≥66% of planned treatments during the DLT observation period or discontinued treatment due to a DLT. Per protocol, DLT outcome analysis did not include Part 3.
Time Frame: Up to approximately 6 weeks
Population: The DLT evaluable population included all participants in Parts 1, 2, 4, and 5 who received at least 66% of all planned treatments during the 6-week DLT observation period or who discontinued treatment due to a DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1:Pembrolizumab 2 mg/kg+dabrafenib150 mg+Trametinib 2 mg; Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg: Participants with BRAF mutant melanoma received 2 mg/kg pembrolizumab administered by IV infusion on Days 1 and 22 Q6W; 150 mg/day total dabrafenib orally, in a divided dose, BID starting on Day 1 and continuing up until study treatment discontinuation; and 2 mg trametinib orally QD starting on Day 1 and continuing up until study treatment discontinuation.
Arm/Group | Part 1:Pembrolizumab 2 mg/kg+dabrafenib150 mg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent
Number analyzed (Participants) | 7 | 3 | 2 | 8 | 2 | 3 | 4 | 5 | 6 | 3 | 12 | 9
Participants | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 2 | 0 | 4 | 2

2. Primary Outcome: Part 2: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator in Participants Without BRAF V600 E or K Mutations
Description: ORR was defined as the percentage of participants without BRAF V600 E or K mutation who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: divided into very good partial response [VGPR; >60% tumor reduction] and moderate partial response [MPR; >30-≤60% tumor reduction]) per RECIST 1.1 as assessed by investigator. The percentage of participants who experienced a CR or PR based on RECIST 1.1 as assessed by investigator were reported.
Time Frame: Up to approximately 85 months
Population: All enrolled participants without BRAF V600 E or K mutations in Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg
Number analyzed (Participants) | 2
Percentage of Participants | 50.0 [1.3 to 98.7]

3. Primary Outcome: Part 5: ORR Per RECIST 1.1 as Assessed by Investigator in Participants Without BRAF V600 E or K Mutations or With Solid Tumors Irrespective of BRAF Status
Description: as for outcome 2
Time Frame: Up to approximately 85 months
Population: All enrolled participants without BRAF V600 E or K mutations in Part 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent
Number analyzed (Participants) | 12 | 9
Percentage of Participants | 0.0 [0.0 to 26.5] | 33.3 [7.5 to 70.1]

4. Primary Outcome: Part 3: Progression-Free Survival (PFS) Per RECIST 1.1 as Assessed by Investigator in Participants With BRAF V600 E or K Mutations
Description: PFS was defined as the time from randomization to the first documented disease progression (PD) or death due to any cause, whichever occurred first, based on RECIST 1.1 by investigator review. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS was analyzed using the Kaplan-Meier method and was reported in months. Statistical analysis used a Cox regression model with treatment as a covariate and stratified by Eastern Cooperative Oncology Group performance status and Lactate Dehydrogenase.
Time Frame: Up to approximately 85 months
Population: All randomized participants with BRAF V600 E or K mutations in Part 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg
Number analyzed (Participants) | 60 | 60
Months | 17.0 [11.3 to NA] — NA = Upper limit for PFS not reached at time of data cut-off due to insufficient number of participants with an event. | 9.9 [6.7 to 15.6]
Statistical Analysis 1: Comparison: Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg vs Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg; Test type: Other; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.29 to 0.74] — Cox regression model

5. Primary Outcome: Parts 1, 2, 4, and 5: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the study drug, was also an AE. The number of participants who experienced an AE was reported. Per protocol, AE outcome analysis did not include Part 3.
Time Frame: Up to approximately 32 months
Population: All participants who received at least one dose of study treatment in Parts 1, 2, 4, and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Pembrolizumab 2 mg/kg+dabrafenib150 mg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent
Number analyzed (Participants) | 7 | 3 | 2 | 8 | 2 | 3 | 4 | 5 | 6 | 3 | 12 | 9
Participants | 7 | 3 | 2 | 8 | 2 | 3 | 4 | 5 | 6 | 3 | 11 | 9

6. Primary Outcome: Parts 1, 2, 4, and 5: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily had to have a causal relationship with this treatment. An AE was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the study drug, was also an AE. The number of participants who discontinued study treatment due to an AE was reported. Per protocol, discontinuation outcome analysis did not include Part 3.
Time Frame: Up to approximately 29 months
Population: All participants who received at least one dose of study treatment in Parts 1, 2, 4, and 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Pembrolizumab 2 mg/kg+dabrafenib150 mg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent
Number analyzed (Participants) | 7 | 3 | 2 | 8 | 2 | 3 | 4 | 5 | 6 | 3 | 12 | 9
Participants | 2 | 2 | 1 | 5 | 2 | 1 | 0 | 4 | 2 | 1 | 2 | 2

7. Secondary Outcome: Part 1: ORR Per RECIST 1.1 as Assessed by Investigator in Participants With BRAF V600 E or K Mutations
Description: ORR was defined as the percentage of participants who had a CR (Disappearance of all target lesions) or a PR (divided into very good partial response [VGPR; >60% tumor reduction] and moderate partial response [MPR; >30-≤60% tumor reduction]) per RECIST 1.1 as assessed by investigator. The percentage of participants who experienced a CR or PR as assessed by the investigator was presented.
Time Frame: Up to approximately 85 months
Population: All enrolled participants with BRAF V600 E or K mutations in Part 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1:Pembrolizumab 2 mg/kg+dabrafenib150 mg+Trametinib 2 mg
Number analyzed (Participants) | 7
Percentage of participants | 57.1 [18.4 to 90.1]

8. Secondary Outcome: Part 2: ORR Per RECIST 1.1 as Assessed by Investigator in Participants With BRAF V600 E or K Mutations
Description: as for outcome 7
Time Frame: Up to approximately 85 months
Population: All enrolled participants with BRAF V600 E or K mutations in Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg
Number analyzed (Participants) | 8
Percentage of Participants | 75.0 [34.9 to 96.8]

9. Secondary Outcome: Part 3: ORR Per RECIST 1.1 as Assessed by Investigator in Participants With BRAF V600 E or K Mutations
Description: as for outcome 7
Time Frame: Up to approximately 85 months
Population: All randomized participants with BRAF V600 E or K mutations in Part 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg
Number analyzed (Participants) | 60 | 60
Percentage of Participants | 65.0 [51.6 to 76.9] | 71.7 [58.6 to 82.5]

10. Secondary Outcome: Part 3: Duration of Response (DOR) Per RECIST 1.1 as Assessed by Investigator in Participants With BRAF V600 E or K Mutations
Description: For participants who demonstrated a confirmed CR (Disappearance of all target lesions) or a confirmed PR (divided by VGPR [>60% tumor reduction] and MPR [>30-≤60% tumor reduction]) per RECIST 1.1 as assessed by the investigator, DOR was defined as the time from first documented evidence of CR or PR until progressive disease (PD). Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. The DOR as assessed by the investigator was analyzed using Kaplan-Meier method and reported in months.
Time Frame: Up to approximately 85 months
Population: All randomized participants with BRAF V600 E or K mutations who had a confirmed CR or PR in Part 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg
Number analyzed (Participants) | 39 | 43
Months | 30.2 [14.1 to NA] — NA = Upper limit for DOR was not reached at time of data cut-off due to insufficient number of responding participants with relapse | 12.1 [6.0 to 15.7]

11. Secondary Outcome: Part 3: Overall Survival (OS) in Participants With BRAF V600 E or K Mutations
Description: OS was defined as the time from randomization to death due to any cause. OS was analyzed using the Kaplan-Meier method and was reported in months. Statistical analysis used a Cox regression model with treatment as a covariate and stratified by Eastern Cooperative Oncology Group performance status and Lactate Dehydrogenase.
Time Frame: Up to approximately 85 months
Population: All randomized participants with BRAF V600 E or K mutations in Part 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg
Number analyzed (Participants) | 60 | 60
Months | 46.3 [23.9 to NA] — NA = Upper limit for OS was not reached at time of data cut-off due to insufficient number of participants with an event | 26.3 [18.2 to 38.6]
Statistical Analysis 1: Comparison: Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg; Test type: Other; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.38 to 0.95] — Cox regression model

12. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab Following Administration of 2 mg/kg Pembrolizumab in Combination With Dabrafenib and/or Trametinib in Participants Pooled From Parts 1 and 2
Description: Cmax was defined as the maximum concentration of pembrolizumab observed after administration of 2 mg/kg pembrolizumab in combination with dabrafenib and/or trametinib. Blood samples were collected at multiple time points to estimate the Cmax of pembrolizumab. All participants who received pembrolizumab from Parts 1 and 2 were handled as a single arm and analyzed as a single study population for this outcome measure since Part 2 was the dose confirmation phase of Part 1. The Cmax of pembrolizumab is presented.
Time Frame: Cycle 1 Day 1: predose, postdose, 24 - 96 hours (hrs) postdose; Cycle 1 Day 22: predose, postdose; Cycle 2 Day 1: predose, postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants pooled from Parts 1 and 2 who received ≥1 dose of 2 mg/kg pembrolizumab and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Pooled Parts 1+2:Pembrolizumab+Dabrafenib+1.5/2 mg Trametinib: Participants pooled from Parts 1 and 2 received 2 mg/kg pembrolizumab in combination with dabrafenib and 2 mg trametinib OR 2 mg/kg pembrolizumab and 1.5 or 2 mg trametinib (without dabrafenib) Q6W continuing up until study treatment discontinuation.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+1.5/2 mg Trametinib
Number analyzed (Participants) | 21
µg/mL | 52.3 (9.9)

13. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab Following Administration of 2 mg/kg Pembrolizumab in Combination With Dabrafenib and Trametinib in Participants From Part 3
Description: Cmax was defined as the maximum concentration of pembrolizumab observed after administration of 2 mg/kg pembrolizumab in combination with dabrafenib and trametinib. Blood samples were collected at multiple time points to estimate the Cmax of pembrolizumab. The Cmax of pembrolizumab is presented.
Time Frame: as for outcome 12
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 2 mg/kg pembrolizumab and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib: Participants received 2 mg/kg pembrolizumab in combination with 150 mg dabrafenib and 2 mg trametinib Q6W continuing up until study treatment discontinuation.
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 58
µg/mL | 48.9 (11.4)

14. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab Following Administration of 200 mg Pembrolizumab in Combination With Trametinib in Participants From Part 4
Description: Cmax was defined as the maximum concentration of pembrolizumab observed after administration of 200 mg pembrolizumab in combination with trametinib. Blood samples were collected at multiple time points to estimate the Cmax of pembrolizumab. The Cmax of pembrolizumab is presented.
Time Frame: Cycle 1 Day 15: predose, postdose, 24 - 96 hrs postdose; Cycle 1 Day 36: predose, postdose; Cycle 2 Day 1: predose, postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 4 who received ≥1 dose of 200 mg pembrolizumab and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Part 4: 200 mg Pembrolizumab+Trametinib: Participants received 2 mg or 1.5 mg trametinib orally QD for 2 or 4 weeks (depending on treatment regimen). Starting with Week 3 or 5 (depending on initial trametinib interval), participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent or concurrent dose schedule of trametinib orally QD continuing up until study treatment discontinuation.
Arm/Group | Part 4: 200 mg Pembrolizumab+Trametinib
Number analyzed (Participants) | 14
µg/mL | 77.8 (16.1)

15. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab Following Administration of 200 mg Pembrolizumab in Combination With Trametinib in Participants From Part 5
Description: as for outcome 14
Time Frame: as for outcome 14
Population: The analysis population consisted of all participants from Part 5 who received ≥1 dose of 200 mg pembrolizumab and who had available data for the analysis of Cmax. There were no participants with data available for the analysis of Cmax in Part 5.
Groups:
- Part 5: 200 mg Pembrolizumab+Trametinib: Participants received 2 mg or 1.5 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent or concurrent dose schedule of trametinib orally QD continuing up until study treatment discontinuation.
Arm/Group | Part 5: 200 mg Pembrolizumab+Trametinib
Number analyzed (Participants) | 0

16. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab Following Administration of 2 mg/kg Pembrolizumab in Combination With Dabrafenib and/or Trametinib in Participants Pooled From Parts 1 and 2
Description: Ctrough was defined as the lowest concentration of pembrolizumab that occurred immediately prior to the next dose of 2 mg/kg pembrolizumab administered in combination with dabrafenib and/or trametinib. Blood samples were collected at multiple time points to estimate the Ctrough of pembrolizumab. All participants who received pembrolizumab from Parts 1 and 2 were handled as a single arm and analyzed as a single study population for this outcome measure since Part 2 was the dose confirmation phase of Part 1. The Ctrough of pembrolizumab is presented.
Time Frame: as for outcome 12
Population: The analysis population consisted of all participants pooled from Parts 1 and 2 who received ≥1 dose of 2 mg/kg pembrolizumab and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+1.5/2 mg Trametinib
Number analyzed (Participants) | 20
µg/mL | 11.2 (2.6)

17. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab Following Administration of 2 mg/kg Pembrolizumab in Combination With Dabrafenib and Trametinib in Participants From Part 3
Description: Ctrough was defined as the lowest concentration of pembrolizumab that occurred immediately prior to the next dose of 2 mg/kg pembrolizumab administered in combination with dabrafenib and trametinib. Blood samples were collected at multiple time points to estimate the Ctrough of pembrolizumab. The Ctrough of pembrolizumab is presented.
Time Frame: as for outcome 12
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 2 mg/kg pembrolizumab and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 49
µg/mL | 10.6 (3.4)

18. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab Following Administration of 200 mg Pembrolizumab in Combination With Trametinib in Participants From Part 4
Description: Ctrough was defined as the lowest concentration of pembrolizumab that occurred immediately prior to the next dose of 200 mg pembrolizumab administered in combination with trametinib. Blood samples were collected at multiple time points to estimate the Ctrough of pembrolizumab. The Ctrough of pembrolizumab is presented.
Time Frame: as for outcome 14
Population: The analysis population consisted of all participants from Part 4 who received ≥1 dose of 200 mg pembrolizumab and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Part 4: 200 mg Pembrolizumab+Trametinib
Number analyzed (Participants) | 15
µg/mL | 17.0 (7.1)

19. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab Following Administration of 200 mg Pembrolizumab in Combination With Trametinib in Participants From Part 5
Description: as for outcome 18
Time Frame: as for outcome 14
Population: The analysis population consisted of all participants from Part 5 who received ≥1 dose of 200 mg pembrolizumab and who had available data for the analysis of Ctrough. There were no participants with data available for the analysis of Ctrough in Part 5.
Arm/Group | Part 5: 200 mg Pembrolizumab+Trametinib
Number analyzed (Participants) | 0

20. Secondary Outcome: Maximum Concentration (Cmax) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With 2 mg/kg Pembrolizumab and 2 mg Trametinib in Participants Pooled From Parts 1 and 2
Description: Cmax was defined as the maximum concentration of dabrafenib observed after administration of 150 mg dabrafenib in combination with 2 mg/kg pembrolizumab and 2 mg trametinib. Blood samples were collected at multiple time points to estimate the Cmax of dabrafenib. All participants who received dabrafenib from Parts 1 and 2 were handled as a single arm and analyzed as a single study population for this outcome measure since Part 2 was the dose confirmation phase of Part 1. The Cmax of dabrafenib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants pooled from Parts 1 and 2 who received ≥1 dose of 150 mg dabrafenib and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pooled Parts 1+2:Pembrolizumab and/or Dabrafenib+2 mg Trametinib: Participants pooled from Parts 1 and 2 received 2 mg/kg pembrolizumab and 150 mg dabrafenib and 2 mg trametinib Q6W continuing up until study treatment discontinuation.
Arm/Group | Pooled Parts 1+2:Pembrolizumab and/or Dabrafenib+2 mg Trametinib
Number analyzed (Participants) | 13
ng/mL | 683 (905)

21. Secondary Outcome: Maximum Concentration (Cmax) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With 2 mg/kg Pembrolizumab and 2 mg Trametinib in Participants From Part 3
Description: Cmax was defined as the maximum concentration of dabrafenib observed after administration of 150 mg dabrafenib in combination with 2 mg/kg pembrolizumab and 2 mg trametinib. Blood samples were collected at multiple time points to estimate the Cmax of dabrafenib. The Cmax of dabrafenib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 150 mg dabrafenib and pembrolizumab and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 53
ng/mL | 643 (643)

22. Secondary Outcome: Maximum Concentration (Cmax) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With Placebo and 2 mg Trametinib in Participants From Part 3
Description: Cmax was defined as the maximum concentration of dabrafenib observed after administration of 150 mg dabrafenib in combination with saline placebo and 2 mg trametinib. Blood samples were collected at multiple time points to estimate the Cmax of dabrafenib. The Cmax of dabrafenib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 150 mg dabrafenib and placebo and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 3: Placebo+Dabrafenib+Trametinib: Participants received saline placebo in combination with 150 mg dabrafenib and 2 mg trametinib Q6W continuing up until study treatment discontinuation.
Arm/Group | Part 3: Placebo+Dabrafenib+Trametinib
Number analyzed (Participants) | 58
ng/mL | 642 (829)

23. Secondary Outcome: Trough Concentration (Ctrough) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With 2 mg/kg Pembrolizumab and 2 mg Trametinib in Participants Pooled From Parts 1 and 2
Description: Ctrough was defined as the lowest concentration of dabrafenib that occurred immediately prior to the next dose of 150 mg dabrafenib administered in combination with 2 mg/kg pembrolizumab and 2 mg trametinib. Blood samples were collected at multiple time points to estimate the Ctrough of dabrafenib. All participants who received dabrafenib from Parts 1 and 2 were handled as a single arm and analyzed as a single study population for this outcome measure since Part 2 was the dose confirmation phase of Part 1. The Ctrough of dabrafenib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants pooled from Parts 1 and 2 who received ≥1 dose of 150 mg dabrafenib and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pooled Parts 1+2:Pembrolizumab and/or Dabrafenib+2 mg Trametinib: Participants pooled from Parts 1 and 2 received 2 mg/kg pembrolizumab in combination with 150 mg dabrafenib and 2 mg trametinib Q6W continuing up until study treatment discontinuation.
Arm/Group | Pooled Parts 1+2:Pembrolizumab and/or Dabrafenib+2 mg Trametinib
Number analyzed (Participants) | 14
ng/mL | 156 (367)

24. Secondary Outcome: Trough Concentration (Ctrough) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With 2 mg/kg Pembrolizumab and 2 mg Trametinib in Participants From Part 3
Description: Ctrough was defined as the lowest concentration of dabrafenib that occurred immediately prior to the next dose of 150 mg dabrafenib administered in combination with 2 mg/kg pembrolizumab and 2 mg trametinib. Blood samples were collected at multiple time points to estimate the Ctrough of dabrafenib. The Ctrough of dabrafenib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 150 mg dabrafenib and pembrolizumab and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 55
ng/mL | 103 (204)

25. Secondary Outcome: Trough Concentration (Ctrough) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With Placebo and 2 mg Trametinib in Participants From Part 3
Description: Ctrough was defined as the lowest concentration of dabrafenib that occurred immediately prior to the next dose of 150 mg dabrafenib administered in combination with saline placebo and 2 mg trametinib. Blood samples were collected at multiple time points to estimate the Ctrough of dabrafenib. The Ctrough of dabrafenib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 150 mg dabrafenib and placebo and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: Placebo+Dabrafenib+Trametinib
Number analyzed (Participants) | 58
ng/mL | 183 (384)

26. Secondary Outcome: Maximum Concentration (Cmax) of Trametinib Following Administration of 2 mg Trametinib in Combination With 2 mg/kg Pembrolizumab and 150 mg Dabrafenib in Participants Pooled From Parts 1 and 2
Description: Cmax was defined as the maximum concentration of trametinib observed after administration of 2 mg trametinib in combination with 2 mg/kg pembrolizumab and 150 mg dabrafenib. Blood samples were collected at multiple time points to estimate the Cmax of trametinib. All participants who received 2 mg trametinib from Parts 1 and 2 were treated as a single arm and analyzed as a single study population for this outcome measure since Part 2 was the dose confirmation phase of Part 1. The Cmax of trametinib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants pooled from Parts 1 and 2 who received ≥1 dose of 2 mg trametinib and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pooled Parts 1+2:Pembrolizumab+Dabrafenib+2 mg Trametinib: Participants pooled from Parts 1 and 2 received 2 mg/kg pembrolizumab in combination with 150 mg dabrafenib and 2 mg trametinib Q6W continuing up until study treatment discontinuation.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+2 mg Trametinib
Number analyzed (Participants) | 13
ng/mL | 19.3 (8.13)

27. Secondary Outcome: Maximum Concentration (Cmax) of Trametinib Following Administration of 1.5 mg Trametinib in Combination With 2 mg/kg Pembrolizumab in Participants Pooled From Parts 1 and 2
Description: Cmax was defined as the maximum concentration of trametinib observed after administration of 1.5 mg trametinib in combination with 2 mg/kg pembrolizumab. Blood samples were collected at multiple time points to estimate the Cmax of trametinib. All participants who received 1.5 mg trametinib from Parts 1 and 2 were treated as a single arm and analyzed as a single study population for this outcome measure since Part 2 was the dose confirmation phase of Part 1. The Cmax of trametinib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants pooled from Parts 1 and 2 who received ≥1 dose of 1.5 mg trametinib and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pooled Parts 1+2:Pembrolizumab+1.5 mg Trametinib: Participants pooled from Parts 1 and 2 received 2 mg/kg pembrolizumab in combination with 1.5 mg trametinib Q6W continuing up until study treatment discontinuation.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 3
ng/mL | 30.3 (17.7)

28. Secondary Outcome: Maximum Concentration (Cmax) of Trametinib Following Administration of 2 mg Trametinib in Combination With 2 mg/kg Pembrolizumab and 150 mg Dabrafenib in Participants From Part 3
Description: Cmax was defined as the maximum concentration of trametinib observed after administration of 2 mg trametinib in combination with 2 mg/kg pembrolizumab and 150 mg dabrafenib. Blood samples were collected at multiple time points to estimate the Cmax of trametinib. The Cmax of trametinib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 2 mg trametinib and pembrolizumab and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 47
ng/mL | 16.3 (6.80)

29. Secondary Outcome: Maximum Concentration (Cmax) of Trametinib Following Administration of 2 mg Trametinib in Combination With Placebo and 150 mg Dabrafenib in Participants From Part 3
Description: Cmax was defined as the maximum concentration of trametinib observed after administration of 2 mg trametinib in combination with saline placebo and 150 mg dabrafenib. Blood samples were collected at multiple time points to estimate the Cmax of trametinib. The Cmax of trametinib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 2 mg trametinib and placebo and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: Placebo+Dabrafenib+Trametinib
Number analyzed (Participants) | 53
ng/mL | 16.2 (6.15)

30. Secondary Outcome: Maximum Concentration (Cmax) of Trametinib Following Administration of 2 mg Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 4
Description: Cmax was defined as the maximum concentration of trametinib observed after administration of 2 mg trametinib in combination with 200 mg pembrolizumab. Blood samples were collected at multiple time points to estimate the Cmax of trametinib. The Cmax of trametinib is presented.
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 4 who received ≥1 dose of 2 mg trametinib and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 4: 200 mg Pembrolizumab+2 mg Trametinib: Participants received 2 mg trametinib orally QD for 2 or 4 weeks (depending on treatment regimen). Starting with Week 3 or 5 (depending on initial trametinib interval), participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent or concurrent dose schedule of 2 mg trametinib orally QD continuing up until study treatment discontinuation.
Arm/Group | Part 4: 200 mg Pembrolizumab+2 mg Trametinib
Number analyzed (Participants) | 4
ng/mL | 18.5 (12.9)

31. Secondary Outcome: Maximum Concentration (Cmax) of Trametinib Following Administration of 1.5 mg Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 4
Description: Cmax was defined as the maximum concentration of trametinib observed after administration of 1.5 mg trametinib in combination with 200 mg pembrolizumab. Blood samples were collected at multiple time points to estimate the Cmax of trametinib. The Cmax of trametinib is presented.
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 4 who received ≥1 dose of 1.5 mg trametinib and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 4: 200 mg Pembrolizumab+1.5 mg Trametinib: Participants received 1.5 mg trametinib orally QD for 2 or 4 weeks (depending on treatment regimen). Starting with Week 3 or 5 (depending on initial trametinib interval), participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent or concurrent dose schedule of 1.5 mg trametinib orally QD continuing up until study treatment discontinuation.
Arm/Group | Part 4: 200 mg Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 7
ng/mL | 16.7 (7.62)

32. Secondary Outcome: Maximum Concentration (Cmax) of Trametinib Following Administration of 2 mg of Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 5
Description: as for outcome 30
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 5 who received ≥1 dose of 2 mg trametinib and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 5: 200 mg Pembrolizumab+2 mg Trametinib: Participants received 2 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent or concurrent dose schedule of 2 mg trametinib orally QD continuing up until study treatment discontinuation.
Arm/Group | Part 5: 200 mg Pembrolizumab+2 mg Trametinib
Number analyzed (Participants) | 3
ng/mL | 7.54 (8.89)

33. Secondary Outcome: Maximum Concentration (Cmax) of Trametinib Following Administration of 1.5 mg of Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 5
Description: as for outcome 31
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 5 who received ≥1 dose of 1.5 mg trametinib and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 5: 200 mg Pembrolizumab+1.5 mg Trametinib: Participants received 1.5 mg trametinib orally QD for 2 weeks. Starting with Week 3, participants received 200 mg pembrolizumab administered by IV infusion on Day 1 Q3W and an intermittent or concurrent dose schedule of 1.5 mg trametinib orally QD continuing up until study treatment discontinuation.
Arm/Group | Part 5: 200 mg Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 8
ng/mL | 14.3 (7.75)

34. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib Following Administration of 2 mg Trametinib in Combination With 2 mg/kg Pembrolizumab and 150 mg Dabrafenib in Participants Pooled From Parts 1 and 2
Description: Ctrough was defined as the lowest concentration of trametinib that occurred immediately prior to the next dose of 2 mg trametinib administered in combination with 2 mg/kg pembrolizumab and 150 mg dabrafenib. Blood samples were collected at multiple time points to estimate the Ctrough of trametinib. All participants who received 2 mg trametinib from Parts 1 and 2 were treated as a single arm and analyzed as a single study population for this outcome measure since Part 2 was the dose confirmation phase of Part 1. The Ctrough of trametinib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants pooled from Parts 1 and 2 who received ≥1 dose of 2 mg trametinib and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+2 mg Trametinib
Number analyzed (Participants) | 14
ng/mL | 13.7 (9.39)

35. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib Following Administration of 1.5 mg Trametinib in Combination With 2 mg/kg Pembrolizumab in Participants Pooled From Parts 1 and 2
Description: Ctrough was defined as the lowest concentration of trametinib that occurred immediately prior to the next dose of 1.5 mg trametinib administered in combination with 2 mg/kg pembrolizumab. Blood samples were collected at multiple time points to estimate the Ctrough of trametinib. All participants who received 1.5 mg trametinib from Parts 1 and 2 were treated as a single arm and analyzed as a single study population for this outcome measure since Part 2 was the dose confirmation phase of Part 1. The Ctrough of trametinib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants pooled from Parts 1 and 2 who received ≥1 dose of 1.5 mg trametinib and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pooled Parts 1+2:Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 3
ng/mL | 20.5 (9.23)

36. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib Following Administration of 2 mg Trametinib in Combination With 2 mg/kg Pembrolizumab and 150 mg Dabrafenib in Participants From Part 3
Description: Ctrough was defined as the lowest concentration of trametinib that occurred immediately prior to the next dose of 2 mg trametinib administered in combination with 2 mg/kg pembrolizumab and 150 mg dabrafenib. Blood samples were collected at multiple time points to estimate the Ctrough of trametinib. The Ctrough of trametinib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 2 mg trametinib and pembrolizumab and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 54
ng/mL | 9.93 (5.48)

37. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib Following Administration of 2 mg Trametinib in Combination With Placebo and 150 mg Dabrafenib in Participants From Part 3
Description: Ctrough was defined as the lowest concentration of trametinib that occurred immediately prior to the next dose of 2 mg trametinib administered in combination with saline placebo and 150 mg dabrafenib. Blood samples were collected at multiple time points to estimate the Ctrough of trametinib. The Ctrough of trametinib is presented.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 3 who received ≥1 dose of 2 mg trametinib and placebo and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: Placebo+Dabrafenib+Trametinib
Number analyzed (Participants) | 58
ng/mL | 10.7 (5.14)

38. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib Following Administration of 2 mg Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 4
Description: Ctrough was defined as the lowest concentration of trametinib that occurred immediately prior to the next dose of 2 mg trametinib administered in combination with 200 mg pembrolizumab. Blood samples were collected at multiple time points to estimate the Ctrough of trametinib. The Ctrough of trametinib is presented.
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 4 who received ≥1 dose of 2 mg trametinib and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 4: 200 mg Pembrolizumab+2 mg Trametinib
Number analyzed (Participants) | 6
ng/mL | 12.3 (9.45)

39. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib Following Administration of 1.5 mg Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 4
Description: Ctrough was defined as the lowest concentration of trametinib that occurred immediately prior to the next dose of 1.5 mg trametinib administered in combination with 200 mg pembrolizumab. Blood samples were collected at multiple time points to estimate the Ctrough of trametinib. The Ctrough of trametinib is presented.
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 4 who received ≥1 dose of 1.5 mg trametinib and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 4: 200 mg Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 7
ng/mL | 8.64 (5.65)

40. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib Following Administration of 2 mg of Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 5
Description: as for outcome 38
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 5 who received ≥1 dose of 2 mg trametinib and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 5: 200 mg Pembrolizumab+2 mg Trametinib
Number analyzed (Participants) | 8
ng/mL | 6.69 (5.9)

41. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib Following Administration of 1.5 mg of Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 5
Description: as for outcome 39
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: The analysis population consisted of all participants from Part 5 who received ≥1 dose of 1.5 mg trametinib and who had available data for the analysis of Ctrough.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 5: 200 mg Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 9
ng/mL | 10.6 (6.79)

42. Secondary Outcome: Clearance (Cl) of Pembrolizumab Following Administration of 2 mg/kg Pembrolizumab in Combination With Dabrafenib and/or Trametinib in Participants Pooled From Parts 1 and 2
Description: Blood samples were to be collected at pre-specified time points for analysis of the Cl of pembrolizumab, defined as the volume of plasma from which pembrolizumab is eliminated per unit time following pembrolizumab administration. This analysis was not performed.
Time Frame: as for outcome 12
Population: As specified by the protocol, the Cl of pembrolizumab was only to be analyzed if required and no data were collected since, by the time of final analysis, pembrolizumab pharmacokinetics (PK) in melanoma participants had been well characterized and found to be consistent with the overall clinical pharmacology of pembrolizumab characterized across indications.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+1.5/2 mg Trametinib
Number analyzed (Participants) | 0

43. Secondary Outcome: Clearance (Cl) of Pembrolizumab Following Administration of 2 mg/kg Pembrolizumab in Combination With Dabrafenib and Trametinib in Participants From Part 3
Description: as for outcome 42
Time Frame: as for outcome 12
Population: as for outcome 42
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

44. Secondary Outcome: Clearance (Cl) of Pembrolizumab Following Administration of 200 mg Pembrolizumab in Combination With Trametinib in Participants From Part 4
Description: as for outcome 42
Time Frame: as for outcome 14
Population: as for outcome 42
Arm/Group | Part 4: 200 mg Pembrolizumab+Trametinib
Number analyzed (Participants) | 0

45. Secondary Outcome: Clearance (Cl) of Pembrolizumab Following Administration of 200 mg Pembrolizumab in Combination With Trametinib in Participants From Part 5
Description: as for outcome 42
Time Frame: as for outcome 14
Population: as for outcome 42
Arm/Group | Part 5: 200 mg Pembrolizumab+Trametinib
Number analyzed (Participants) | 0

46. Secondary Outcome: Clearance (Cl) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With 2 mg/kg Pembrolizumab and 2 mg Trametinib in Participants Pooled From Parts 1 and 2
Description: Blood samples were to be collected at pre-specified time points for analysis of the Cl of dabrafenib, defined as the volume of plasma from which dabrafenib is eliminated per unit time following dabrafenib administration. This analysis was not performed.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: As specified by the protocol, the Cl of dabrafenib was only to be analyzed if required and no data were collected since, by the time of final analysis, dabrafenib pharmacokinetics (PK) in melanoma participants had been well characterized and found to be consistent with the overall clinical pharmacology of dabrafenib characterized across indications.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+2 mg Trametinib
Number analyzed (Participants) | 0

47. Secondary Outcome: Clearance (Cl) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With 2 mg/kg Pembrolizumab and 2 mg Trametinib in Participants From Part 3
Description: as for outcome 46
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 46
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

48. Secondary Outcome: Clearance (Cl) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With Placebo and 2 mg Trametinib in Participants From Part 3
Description: as for outcome 46
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 46
Arm/Group | Part 3: Placebo+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

49. Secondary Outcome: Clearance (Cl) of Trametinib Following Administration of 2 mg Trametinib in Combination With 2 mg/kg Pembrolizumab and 150 mg Dabrafenib in Participants Pooled From Parts 1 and 2
Description: Blood samples were to be collected at pre-specified time points for analysis of the Cl of trametinib, defined as the volume of plasma from which trametinib is eliminated per unit time following trametinib administration. This analysis was not performed.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: As specified by the protocol, the Cl of trametinib was only to be analyzed if required and no data were collected since, by the time of final analysis, trametinib pharmacokinetics (PK) in melanoma participants had been well characterized and found to be consistent with the overall clinical pharmacology of trametinib characterized across indications.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+2 mg Trametinib
Number analyzed (Participants) | 0

50. Secondary Outcome: Clearance (Cl) of Trametinib Following Administration of 1.5 mg Trametinib in Combination With 2 mg/kg Pembrolizumab in Participants Pooled From Parts 1 and 2
Description: as for outcome 49
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 49
Arm/Group | Pooled Parts 1+2:Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 0

51. Secondary Outcome: Clearance (Cl) of Trametinib Following Administration of 2 mg Trametinib in Combination With 2 mg/kg Pembrolizumab and 150 mg Dabrafenib in Participants From Part 3
Description: as for outcome 49
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 49
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

52. Secondary Outcome: Clearance (Cl) of Trametinib Following Administration of 2 mg Trametinib in Combination With Placebo and 150 mg Dabrafenib in Participants From Part 3
Description: as for outcome 49
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 49
Arm/Group | Part 3: Placebo+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

53. Secondary Outcome: Clearance (Cl) of Trametinib Following Administration of 2 mg Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 4
Description: as for outcome 49
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 49
Arm/Group | Part 4: 200 mg Pembrolizumab+2 mg Trametinib
Number analyzed (Participants) | 0

54. Secondary Outcome: Clearance (Cl) of Trametinib Following Administration of 1.5 mg Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 4
Description: as for outcome 49
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 49
Arm/Group | Part 4: 200 mg Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 0

55. Secondary Outcome: Clearance (Cl) of Trametinib Following Administration of 2 mg of Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 5
Description: as for outcome 49
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 49
Arm/Group | Part 5: 200 mg Pembrolizumab+2 mg Trametinib
Number analyzed (Participants) | 0

56. Secondary Outcome: Clearance (Cl) of Trametinib Following Administration of 1.5 mg of Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 5
Description: as for outcome 49
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 49
Arm/Group | Part 5: 200 mg Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 0

57. Secondary Outcome: Volume of Distribution (Vc) of Pembrolizumab Following Administration of 2 mg/kg Pembrolizumab in Combination With Dabrafenib and/or Trametinib in Participants Pooled From Parts 1 and 2
Description: Blood samples were to be collected at pre-specified time points for analysis of the Vc of pembrolizumab, defined as the theoretical volume that would be necessary to contain the total amount of administered pembrolizumab at the same concentration that it is observed in the blood plasma. This analysis was not performed.
Time Frame: as for outcome 12
Population: As specified by the protocol, the Vc of pembrolizumab was only to be analyzed if required and no data were collected since, by the time of final analysis, pembrolizumab pharmacokinetics (PK) in melanoma participants had been well characterized and found to be consistent with the overall clinical pharmacology of pembrolizumab characterized across indications.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+1.5/2 mg Trametinib
Number analyzed (Participants) | 0

58. Secondary Outcome: Volume of Distribution (Vc) of Pembrolizumab Following Administration of 2 mg/kg Pembrolizumab in Combination With Dabrafenib and Trametinib in Participants From Part 3
Description: as for outcome 57
Time Frame: as for outcome 12
Population: as for outcome 57
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

59. Secondary Outcome: Volume of Distribution (Vc) of Pembrolizumab Following Administration of 200 mg Pembrolizumab in Combination With Trametinib in Participants From Part 4
Description: as for outcome 57
Time Frame: as for outcome 14
Population: as for outcome 57
Arm/Group | Part 4: 200 mg Pembrolizumab+Trametinib
Number analyzed (Participants) | 0

60. Secondary Outcome: Volume of Distribution (Vc) of Pembrolizumab Following Administration of 200 mg Pembrolizumab in Combination With Trametinib in Participants From Part 5
Description: as for outcome 57
Time Frame: as for outcome 14
Population: as for outcome 57
Arm/Group | Part 5: 200 mg Pembrolizumab+Trametinib
Number analyzed (Participants) | 0

61. Secondary Outcome: Volume of Distribution (Vc) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With 2 mg/kg Pembrolizumab and 2 mg Trametinib in Participants Pooled From Parts 1 and 2
Description: Blood samples were to be collected at pre-specified time points for analysis of the Vc of dabrafenib, defined as the theoretical volume that would be necessary to contain the total amount of administered dabrafenib at the same concentration that it is observed in the blood plasma. This analysis was not performed.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: As specified by the protocol, the Vc of dabrafenib was only to be analyzed if required and no data were collected since, by the time of final analysis, dabrafenib pharmacokinetics (PK) in melanoma participants had been well characterized and found to be consistent with the overall clinical pharmacology of dabrafenib characterized across indications.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+2 mg Trametinib
Number analyzed (Participants) | 0

62. Secondary Outcome: Volume of Distribution (Vc) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With 2 mg/kg Pembrolizumab and 2 mg Trametinib in Participants From Part 3
Description: as for outcome 61
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 61
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

63. Secondary Outcome: Volume of Distribution (Vc) of Dabrafenib Following Administration of 150 mg Dabrafenib in Combination With Placebo and 2 mg Trametinib in Participants From Part 3
Description: as for outcome 61
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 61
Arm/Group | Part 3: Placebo+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

64. Secondary Outcome: Volume of Distribution (Vc) of Trametinib Following Administration of 2 mg Trametinib in Combination With 2 mg/kg Pembrolizumab and 150 mg Dabrafenib in Participants Pooled From Parts 1 and 2
Description: Blood samples were to be collected at pre-specified time points for analysis of the Vc of trametinib, defined as the theoretical volume that would be necessary to contain the total amount of administered trametinib at the same concentration that it is observed in the blood plasma. This analysis was not performed.
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: As specified by the protocol, the Vc of trametinib was only to be analyzed if required and no data were collected since, by the time of final analysis, trametinib pharmacokinetics (PK) in melanoma participants had been well characterized and found to be consistent with the overall clinical pharmacology of trametinib characterized across indications.
Arm/Group | Pooled Parts 1+2:Pembrolizumab+Dabrafenib+2 mg Trametinib
Number analyzed (Participants) | 0

65. Secondary Outcome: Volume of Distribution (Vc) of Trametinib Following Administration of 1.5 mg Trametinib in Combination With 2 mg/kg Pembrolizumab in Participants Pooled From Parts 1 and 2
Description: as for outcome 64
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 64
Arm/Group | Pooled Parts 1+2:Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 0

66. Secondary Outcome: Volume of Distribution (Vc) of Trametinib Following Administration of 2 mg Trametinib in Combination With 2 mg/kg Pembrolizumab and 150 mg Dabrafenib in Participants From Part 3
Description: as for outcome 64
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 64
Arm/Group | Part 3: 2 mg/kg Pembrolizumab+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

67. Secondary Outcome: Volume of Distribution (Vc) of Trametinib Following Administration of 2 mg Trametinib in Combination With Placebo and 150 mg Dabrafenib in Participants From Part 3
Description: as for outcome 64
Time Frame: Cycle 1 Day 22: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 64
Arm/Group | Part 3: Placebo+Dabrafenib+Trametinib
Number analyzed (Participants) | 0

68. Secondary Outcome: Volume of Distribution (Vc) of Trametinib Following Administration of 2 mg Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 4
Description: as for outcome 64
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 64
Arm/Group | Part 4: 200 mg Pembrolizumab+2 mg Trametinib
Number analyzed (Participants) | 0

69. Secondary Outcome: Volume of Distribution (Vc) of Trametinib Following Administration of 1.5 mg Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 4
Description: as for outcome 64
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 64
Arm/Group | Part 4: 200 mg Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 0

70. Secondary Outcome: Volume of Distribution (Vc) of Trametinib Following Administration of 2 mg of Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 5
Description: as for outcome 64
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 64
Arm/Group | Part 5: 200 mg Pembrolizumab+2 mg Trametinib
Number analyzed (Participants) | 0

71. Secondary Outcome: Volume of Distribution (Vc) of Trametinib Following Administration of 1.5 mg of Trametinib in Combination With 200 mg Pembrolizumab in Participants From Part 5
Description: as for outcome 64
Time Frame: Cycle 1 Day 36: predose, postdose, 4 - 6 hrs postdose. Each cycle is a 21-day cycle.
Population: as for outcome 64
Arm/Group | Part 5: 200 mg Pembrolizumab+1.5 mg Trametinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 85 months
Description: All-cause mortality=all randomized participants and adverse events (AE)=all participants who received ≥1 dose of treatment. Per protocol, disease progression was not considered an AE unless related to treatment. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression, malignant neoplasm progression, and disease progression not related to treatment were excluded.
Arm/Group | Part 1:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 2 mg | Part 1:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg | Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent
All-Cause Mortality (participants affected / at risk) | 4/7 | 1/3 | 1/2 | 3/8 | 2/2 | 31/60 | 45/60 | 2/3 | 3/4 | 4/5 | 5/6 | 3/3 | 11/12 | 7/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/3 | 1/2 | 3/8 | 1/2 | 36/60 | 20/60 | 1/3 | 1/4 | 4/5 | 4/6 | 1/3 | 4/12 | 2/9
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 2/2 | 8/8 | 2/2 | 60/60 | 58/60 | 3/3 | 4/4 | 5/5 | 6/6 | 3/3 | 11/12 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg (N=7) | Part 1:Pembrolizumab 2 mg/kg+Trametinib 2 mg (N=3) | Part 1:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg (N=2) | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg (N=8) | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg (N=2) | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg (N=60) | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg (N=60) | Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg (N=3) | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg (N=4) | Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg (N=5) | Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent (N=6) | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent (N=3) | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg (N=12) | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discoloured vomit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (9) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute motor axonal neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg (N=7) | Part 1:Pembrolizumab 2 mg/kg+Trametinib 2 mg (N=3) | Part 1:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg (N=2) | Part 2:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg (N=8) | Part 2:Pembrolizumab 2 mg/kg+Trametinib 1.5 mg (N=2) | Part 3:Pembrolizumab 2 mg/kg+Dabrafenib 150 mg+Trametinib 2 mg (N=60) | Part 3:Placebo+Dabrafenib 150 mg+Trametinib 2 mg (N=60) | Part 4:4 Weeks Trametinib (Tra) 2mg; Pembrolizumab+Tra 2mg (N=3) | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg (N=4) | Part 4:4 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg (N=5) | Part 4:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent (N=6) | Part 4:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg Intermittent (N=3) | Part 5:2 Weeks Tra 1.5mg; Pembrolizumab+Tra 1.5mg (N=12) | Part 5:2 Weeks Tra 2mg; Pembrolizumab+Tra 2mg Intermittent (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (13) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 6 (6) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chorioretinal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid rash (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 1 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous adhesions (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (7) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 3 (4)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (3) | 2 (2) | 1 (1) | 0 (0) | 5 (7) | 7 (7) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (9) | 2 (6) | 2 (5) | 6 (8) | 0 (0) | 28 (90) | 17 (29) | 3 (4) | 2 (3) | 2 (5) | 5 (15) | 1 (1) | 5 (12) | 5 (11)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (7) | 1 (2) | 5 (9) | 0 (0) | 23 (46) | 28 (47) | 0 (0) | 1 (1) | 3 (3) | 3 (5) | 2 (2) | 3 (4) | 2 (2)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (7) | 0 (0) | 22 (55) | 17 (29) | 0 (0) | 1 (1) | 2 (3) | 3 (8) | 1 (1) | 2 (2) | 2 (3)
Asthenia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 19 (33) | 11 (14) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 6 (21) | 2 (2) | 0 (0) | 6 (12) | 0 (0) | 21 (59) | 23 (51) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 1 (1) | 2 (2) | 6 (10) | 1 (2) | 22 (37) | 25 (41) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 3 (3)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (15) | 8 (12) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (8) | 0 (0) | 2 (2) | 2 (2) | 10 (13) | 5 (5) | 1 (2) | 1 (1) | 2 (2) | 3 (3) | 1 (2) | 4 (5) | 4 (4)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 7 (23) | 2 (3) | 0 (0) | 8 (25) | 0 (0) | 50 (262) | 41 (118) | 1 (2) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 7 (14) | 3 (4)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 6 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 6 (9) | 5 (7) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 8 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 11 (15) | 11 (12) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 6 (8) | 3 (5)
Amylase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 12 (17) | 12 (14) | 0 (0) | 3 (3) | 2 (4) | 3 (4) | 0 (0) | 6 (10) | 5 (8)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 10 (18) | 12 (16) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (9) | 6 (9) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 5 (8) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 10 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (7) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 13 (17) | 11 (11) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (2) | 1 (1) | 4 (12) | 0 (0) | 24 (54) | 17 (34) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 8 (9) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (12) | 0 (0) | 16 (23) | 10 (17) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 7 (11) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Winged scapula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 7 (8) | 8 (10) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
External compression headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 2 (4) | 0 (0) | 4 (6) | 0 (0) | 18 (29) | 13 (23) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 4 (4) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 10 (17) | 12 (12) | 1 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 4 (6) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (2) | 1 (1) | 9 (11) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 5 (5) | 8 (12) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 0 (0) | 4 (5) | 0 (0) | 9 (9) | 4 (4) | 3 (4) | 3 (7) | 2 (5) | 5 (6) | 1 (1) | 3 (4) | 6 (7)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 7 (10) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 7 (12) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 6 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (6) | 3 (5) | 1 (1) | 2 (2) | 1 (2) | 10 (17) | 9 (12) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 2 (3) | 6 (10) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (8) | 2 (5) | 1 (3) | 4 (5) | 1 (1) | 27 (50) | 18 (24) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 3 (5) | 6 (11) | 3 (6)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash follicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (9) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 3 (4) | 0 (0) | 2 (2) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 12 (18) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (12) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 10 (13) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT02130466/Prot_SAP_000.pdf